CLINICAL TRIAL: NCT04575688
Title: A Randomized Controlled Trial Comparing a Periarticular Injection to a Popliteal Block for Pain Control in Ankle/Hindfoot Osteotomy or Fusion and Ankle Fractures
Brief Title: Periarticular Injection Versus Popliteal Block
Acronym: PvP
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Campbell Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-06453-FB
Record Dates: First submitted 2020-09-23; First posted 2020-10-05 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Foot Surgery; Ankle Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Periarticular Injection (Active Comparator): Subjects undergoing hindfoot osteotomy or fusion, ankle osteotomy or fusion, or ankle fracture repair will recieve a periarticular injection by the surgeon using 10 milliliters of Exparel mixed with 10 milliliters of bupivicaine 0.5 percent at the end of the procedure.
  Interventions: Drug: Exparel
- Popliteal Block (Active Comparator): Subjects undergoing hindfoot osteotomy or fusion, ankle osteotomy or fusion, or ankle fracture repair will recieve a popliteal block by the anesthesiologist using 30 milliliters of bupivicaine 0.5 percent in the pre-operative area, prior to surgery, using an ultrasound machine for guidance.
  Interventions: Drug: Bupivicaine

INTERVENTIONS:
Drug: Exparel — Exparel will be administered by periarticular injection to patients undergoing hindfoot osteotomy or fusion, ankle osteotomy or fusion, or ankle fracture repair.
  Other Names: Periarticular Injection
  Arms: Periarticular Injection
Drug: Bupivicaine — Bupivicaine will be administered by popliteal block to patients undergoing hindfoot osteotomy or fusion, ankle osteotomy or fusion, or ankle fracture repair.
  Other Names: Peripheral Nerve Injection
  Arms: Popliteal Block

SUMMARY:
This study aims to determine the effectiveness and safety of two standard of care perioperative procedures for controlling pain following ankle and hindfoot osteotomy or fusion or ankle fracture repair.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled research study of two perioperative standards of care for managing post operative pain. The first standard of care procedure is the periarticular injection; the second is the popiteal block.

ELIGIBILITY:
Inclusion Criteria:

* Ankle or hindfoot osteotomy or ankle fracture repair
* Surgery scheduled at Campbell Surgery Center (1410 Brierbrook Road, Germantown, TN 38138)
* 18-80 years of age
* ASA I-III with medical clearances as needed
* Fluent ub verbal and written English
* Willing and able to comply with study instruction and commit to all follow-up visits for theduration of the study
* Willing and able to provide written consent

Exclusion Criteria:

* Diagnosed with chronic pain syndrome
* History of allergic reactions to lidocaine, marcaine, Experal, bupivicaine, or other injectable anesthetic agents
* Injury associated with workers' compensation
* Surgery to be performed at a hospital
* Diagnosed with peripheral neuropathy
* Hbg A1C is > 7 mg/dl in diabetic patients only
* Long term (chronic) preoperative narcotic usage

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-13 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Score | Postoperative hour 3
  Patient reported pain score from zero to ten where zero is no pain and ten is the most pain
Evidence of motor block | Postoperative hour 3
  Patient reported yes/no answer to survey question: "Are you able to wiggle your toes?"
Visual Analog Score | Postoperative hour 6
  Patient reported pain score from zero to ten where zero is no pain and ten is the most pain
Visual Analog Score | Postoperative hour 12
  Patient reported pain score from zero to ten where zero is no pain and ten is the most pain
Visual Analog Score | Postoperative hour 24
  Patient reported pain score from zero to ten where zero is no pain and ten is the most pain
Visual Analog Score | Postoperative hour 36
  Patient reported pain score from zero to ten where zero is no pain and ten is the most pain
Visual Analog Score | Postoperative hour 48
  Patient reported pain score from zero to ten where zero is no pain and ten is the most pain
Visual Analog Score | Postoperative hour 72
  Patient reported pain score from zero to ten where zero is no pain and ten is the most pain
Visual Analog Score | Postoperative week 2
  Patient reported pain score from zero to ten where zero is no pain and ten is the most pain
Visual Analog Score | Postoperative week 4-6
  Patient reported pain score from zero to ten where zero is no pain and ten is the most pain
Visual Analog Score | Postoperative week 12
  Patient reported pain score from zero to ten where zero is no pain and ten is the most pain

SECONDARY OUTCOMES:
Document pain medication prescribed immediately after surgery | Immediately after surgery
  Pain medication prescribed immediately after the surgery will be documented in the research record. This is a descriptive data point to capture the incidence of narcotics prescribed immediately after surgery, to include opiate name, dose, and number of pills prescribed.
Satisfaction with pain control: survey question | Postoperative week 2
  Patient reported 7-point Likert scale answer to survey question: "How satisfied are you with your pain control?" 1 = very dissatisfied, 2 = dissatisfied, 3 = moderately dissatisfied, 4 = neutral, 5 = moderately satisfied, 6 = satisfied, 7 = very satisfied.
Neuralgia symptoms: survey question | Postoperative week two
  Patient reported yes/no answer to survey question: "Have you had any signs of neuralgia, such as persistent numbness, tingling, or increased sensitivity in your foot or ankle that you feel is not at the surgical location?" 1 = yes, I have had signs of neuralgia; 2 = no, I have not had signs of neuralgia.
Pill count | Postoperative week 2
  Patient reported fill-in-the-blank answer to survey question: "Total number of pain pills taken during this time."
Document pain medication prescribed at postoperative week 2 | Postoperative week 2
  Pain medication prescribed at postoperative week 2 will be documented in the research record. This is a descriptive data point to capture the incidence of narcotics prescribed at postoperative week 2, to include opiate name, dose, and number of pills prescribed.
Satisfaction with pain control: survey question | Postoperative week 6
  Patient reported 7-point Likert scale answer to survey question: "How satisfied are you with your pain control?" Patient reported 7-point Likert scale answer to survey question: "How satisfied are you with your pain control?" 1 = very dissatisfied, 2 = dissatisfied, 3 = moderately dissatisfied, 4 = neutral, 5 = moderately satisfied, 6 = satisfied, 7 = very satisfied.
Neuralgia symptoms: survey question | Postoperative week 6
  Patient reported yes/no answer to survey question: "Have you had any signs of neuralgia, such as persistent numbness, tingling, or increased sensitivity in your foot or ankle that you feel is not at the surgical location?" 1 = yes, I have had signs of neuralgia; 2 = no, I have not had signs of neuralgia.
Pill count | Postoperative week 6
  Patient reported fill-in-the-blank answer to survey question: "Total number of pain pills taken during this time."
Document pain medication prescribed at postoperative week 6 | Postoperative week 6
  Pain medication prescribed at postoperative week 6 will be documented in the research record. This is a descriptive data point to capture the incidence of narcotics prescribed at postoperative week 6, to include opiate name, dose, and number of pills prescribed.
Satisfaction with pain control: survey question | Postoperative week 12
  Patient reported 7-point Likert scale answer to survey question: "How satisfied are you with your pain control?" Patient reported 7-point Likert scale answer to survey question: "How satisfied are you with your pain control?" 1 = very dissatisfied, 2 = dissatisfied, 3 = moderately dissatisfied, 4 = neutral, 5 = moderately satisfied, 6 = satisfied, 7 = very satisfied.
Neuralgia symptoms: survey question | Postoperative week 12
  Patient reported yes/no answer to survey question: "Have you had any signs of neuralgia, such as persistent numbness, tingling, or increased sensitivity in your foot or ankle that you feel is not at the surgical location?" 1 = yes, I have had signs of neuralgia; 2 = no, I have not had signs of neuralgia.
Pill count | Postoperative week 12
  Patient reported fill-in-the-blank answer to survey question: "Total number of pain pills taken during this time."
Document pain medication prescribed at postoperative week 12 | Postoperative week 12
  Pain medication prescribed at postoperative week 12 will be documented in the research record. This is a descriptive data point to capture the incidence of narcotics prescribed at postoperative week 12, to include opiate name, dose, and number of pills prescribed.

CONTACTS AND LOCATIONS:
Overall Officials: Garnett A Murphy, MD, Principal Investigator — Campbell Clinic
Locations (1):
- A, Germantown, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No